CLINICAL TRIAL: NCT03316950
Title: A Randomized, Placebo-Controlled Trial Evaluating Radiofrequency and Hybrid Fractional Laser for Vaginal Rejuvenation
Brief Title: Radiofrequency and Hybrid Fractional Laser for Vaginal Rejuvenation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: American Society for Aesthetic Plastic Surgery (Other)
Responsible Party: Principal Investigator, Jeffrey M. Kenkel, Chair, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU 012017-006
Record Dates: First submitted 2017-10-17; First posted 2017-10-23 (Actual); Results first posted 2023-01-04 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2022-12

CONDITIONS: Vaginal Atrophy
Keywords: postmenopause; rejuvenation; radiofrequency; diva

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- IntraGen RF (Experimental): Patients will undergo treatment with radiofrequency device, using the device's standard protocol. Patients will have 3 treatments space one month apart. Each treatment will be a total of 20 minutes for internal treatment only. Prior to treatment, the Zimmern probe will be used to measure vaginal wall elasticity and a 0.33mm biopsy will be taken. At each visit, the Zimmern probe will be used. Biopsies will be taken 3 months after final treatment.
  Interventions: Device: IntraGen RF
- DiVA (Experimental): Patients randomized into the DiVA treatment group will receive treatment per DiVA protocol. Patients will have a total of 3 treatments, space 1 month apart. Each treatment will last approximately 10 minutes. Prior to treatment, the Zimmern probe will be used to measure vaginal wall elasticity and a 0.33mm biopsy will be taken. At each visit, the Zimmern probe will be used. Biopsies will be taken 3 months after final treatment.
  Interventions: Device: DiVA
- Placebo Arm (Sham Comparator): Patients randomized into the Placebo arm will include participants from the DiVa PlaceboGroup and IntraGen Placebo Group combined and will receive treatment based on the DiVA Sham and IntraGen Sham protocols.
  DiVa Placebo: patients will undergo a three-part placebo treatment, spaced 1 month apart (+/- 10 days) of the vulvovaginal area. The vaginal HFL handpiece will be inserted into the vaginal canal but sub-therapeutic energy will not be delivered to the tissue.
  IntraGen Placebo: patients will undergo a three-part placebo treatment, space 1 month apart (+/- 10 days) of the vulvovaginal area. This will be achieved through application of the probe, but with applying sub-therapeutic energy to the tissue.
  Interventions: Device: Placebo (DIVA/IntraGen combined)
- Dual Treatment (Experimental): Patients previously randomized into the DiVA Sham and IntraGen Sham groups will be placed in the Dual Treatment group. Patients will have a total of 3 dual treatments, spaced 1 month apart. Each treatment will last approximately 20 minutes. Prior to dual treatments, the Zimmern probe will be used to measure vaginal wall elasticity and a 0.33mm biopsy will be taken. At each visit, the Zimmern probe will be used. Biopsies will be taken at follow up visits.
  Interventions: Device: IntraGen RF; Device: DiVA

INTERVENTIONS:
Device: IntraGen RF — IntraGen is a radiofrequency vaginal rejuvenation device FDA approved for use in dermatological and general surgical procedures for electrocoagulation and hemostasis. The hand piece is a disposable monopolar applicator that is used to apply energy internally and externally.
  Arms: Dual Treatment; IntraGen RF
Device: DiVA — DiVA device utilizes a hybrid fractional laser technology in a wand hand piece. The hand piece is covered by a single use strengthened quartz dilator that allows the hand piece to rotate and provide treatment in a uniform manner.
  Arms: DiVA; Dual Treatment
Device: Placebo (DIVA/IntraGen combined) — (DIVA/IntraGen combined) IntraGen RF: IntraGen is a radiofrequency vaginal rejuvenation device FDA approved for use in dermatological and general surgical procedures for electrocoagulation and hemostasis. The hand piece is a disposable monopolar applicator that is used to apply energy internally and externally.
  DiVA: DiVA device utilizes a hybrid fractional laser technology in a wand hand piece. The hand piece is covered by a single use strengthened quartz dilator that allows the hand piece to rotate and provide treatment in a uniform manner.
  Arms: Placebo Arm

SUMMARY:
This is a single-center, randomized, prospective study designed to evaluate the efficacy of radiofrequency and hybrid fractional laser for vaginal rejuvenation. 120 subjects will be screened with 100 undergoing a three-part treatment of the vulvovaginal area IntraGen RF unit, IntraGen RF unit placebo, DiVa HFL unit, or DiVa HFL unit placebo. These treatments will be spaced one month apart and last about 25 minutes each. Each subject will be screened, undergo testing at baseline, and will be followed conservatively with no further therapy until they reach 6 months after the initiation of the designated treatment. At that time, all subjects will undergo subjective and objective testing. Those in the treatment group will be followed to 9 and 12 months after the initiation of treatment with appropriate analysis. Those in the placebo group will be provided a three-part treatment of the vulvovaginal area with the IntraGen RF unit and DiVA HFL unit. These treatments will be spaced one month apart and last about 25 minutes each. Six months after receiving three treatments of the dual therapy these patients will undergo subjective and objective testing. The primary outcome measure is improvement in vulvovaginal symptoms measured by the validated Vulvovaginal Symptoms Questionnaire. Data obtained from each investigation will be recorded in a password-protected digital spreadsheet, REDCap database and descriptive statistics will be obtained.

DETAILED DESCRIPTION:
Vaginal rejuvenation is a catch-all term of trendy procedures which claim to provide relief of many issues affecting women's health, ranging from postmenopausal vulvovaginal symptoms (i.e. dryness, burning, itching), stress urinary incontinence, sexual dysfunction or discomfort, vaginal laxity, and labial appearance, amongst others2,3. Several companies have emerged with non-invasive or minimally-invasive technologies to alleviate these conditions which operate by radiofrequency delivery (IntraGen by Jeisys), Hybrid Fractional Laser (diVa by Sciton), or fractional CO2 laser (Mona Lisa Touch by Cynosure and Femi Lift by Alma Laser)4.

All of these technologies work theoretically by remodeling extracellular matrix configuration. It is of important note that radiofrequency therapies are typically delivered at 45-55 degrees Celsius in the tissues whereas the laser based products heat up to 60-70 degrees Celsius5. It is believed that "neocollagenesis" may only start if the temperatures are high enough and that such changes in the collagen matrix of the vagina could lead to durable vaginal wall changes. Sciton's diVa is hybrid fractional laser with wavelengths of 2940 nm and 1470 nm for ablation and coagulation, respectively, to treat vaginal tissue6. It is not known whether the changes experienced by patients are due to the reconfiguration of the extracellular matrix (ECM) deep in the vaginal wall or related to the acute swelling and inflammatory processes that occur at the surface of the vagina after these rejuvenation procedures.

The early anecdotal success reported on some user websites might be attributable to surface changes that may not be lasting or to possibly more lasting deeper muscular vaginal wall changes, which may or may not be beneficial. Based on the answer to this first set of questions, we might possibly surmise how such changes will ultimately improve vaginal dryness and/or stress urinary incontinence complaints.

An overriding question and concern is: Assuming these treatments induce collagen changes in the vagina, is it safe to induce such changes? If changes occur, are they long lasting? Can it age the vagina instead of making it "younger"? What are the long-term effects of doing so? Is tissue tightening really scar formation that may be deleterious in the future? The histological, genetic and dynamic changes following vaginal rejuvenation have never been studied.

ELIGIBILITY:
Inclusion Criteria:

* Women should be between 40 and 65 years of age
* Women should be post-menopausal
* Women should be amenorrheic for at least 12 months
* Postmenopausal women presenting with one or more of the following:
* Vulvar itching
* Vulvar burning or stinging
* Vulvar pain
* Vulvar irritation
* Vulvar dryness
* Discharge from subject's vulva or vagina
* Odor from subject's vulva or vagina

Exclusion Criteria:

* Unable to commit to future appointments within one year
* Planning on moving away from Dallas within one year
* History of other energy-based vaginal therapy within one year
* Vaginal hormone replacement therapy must have a one month washout period prior to treatment and discontinued use for duration of study, systemic replacement is not excluded
* Prior labiaplasty, or vaginal injections of fat or fillers within 6 months
* Prior anti-incontinence surgery in the last 12 months
* Urinary incontinence requiring more than 2 pads/day
* Clinically significant pelvic organ prolapse (POP)
* Urinary tract infection in the past 3 months
* Unstable diabetes
* Ongoing chemotherapy
* Immunodeficiency status (steroid intake, ongoing chemotherapy)
* Diffuse pain syndrome or chronic pain requiring daily narcotics
* Chronic vaginitis including bacterial vaginosis, HPV, herpes, or other active STI
* Recent abnormal Papanicolaou test result
* Recent abnormal pelvic exam (i.e. concerning lesions)
* Vulvar dermatologic pathology requiring local steroid use
* Undiagnosed abnormal genital bleeding
* If less than two years postmenopausal, not using a medically approved method of contraception (i.e. oral, transdermal, implanted contraceptives, intrauterine device, diaphragm, condom, etc.)
* Pregnancy
* History of genital fistula or a thin rectovaginal septum
* Uncontrolled psychiatric conditions (well-controlled depression/anxiety is not excluded)
* Body Mass Index > 35
* Actively participating in or planning on participating in pelvic floor muscle strengthening exercise
* Presence of pacemaker, AICD, or other electrical health maintenance device

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2021-04-08 (Actual); Study Completion 2021-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Kenkel, MD, Principal Investigator — Chair & Professor
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alinsod RM. Transcutaneous temperature controlled radiofrequency for orgasmic dysfunction. Lasers Surg Med. 2016 Sep;48(7):641-5. doi: 10.1002/lsm.22537. Epub 2016 May 19. PMID 27197701
- [Background] Millheiser LS, Pauls RN, Herbst SJ, Chen BH. Radiofrequency treatment of vaginal laxity after vaginal delivery: nonsurgical vaginal tightening. J Sex Med. 2010 Sep;7(9):3088-95. doi: 10.1111/j.1743-6109.2010.01910.x. PMID 20584127
- [Background] Sekiguchi Y, Utsugisawa Y, Azekosi Y, Kinjo M, Song M, Kubota Y, Kingsberg SA, Krychman ML. Laxity of the vaginal introitus after childbirth: nonsurgical outpatient procedure for vaginal tissue restoration and improved sexual satisfaction using low-energy radiofrequency thermal therapy. J Womens Health (Larchmt). 2013 Sep;22(9):775-81. doi: 10.1089/jwh.2012.4123. Epub 2013 Aug 16. PMID 23952177
- [Background] Zerbinati N, Serati M, Origoni M, Candiani M, Iannitti T, Salvatore S, Marotta F, Calligaro A. Microscopic and ultrastructural modifications of postmenopausal atrophic vaginal mucosa after fractional carbon dioxide laser treatment. Lasers Med Sci. 2015 Jan;30(1):429-36. doi: 10.1007/s10103-014-1677-2. Epub 2014 Nov 20. PMID 25410301
- [Background] Paul M, Blugerman G, Kreindel M, Mulholland RS. Three-dimensional radiofrequency tissue tightening: a proposed mechanism and applications for body contouring. Aesthetic Plast Surg. 2011 Feb;35(1):87-95. doi: 10.1007/s00266-010-9564-0. Epub 2010 Sep 11. PMID 20835826
- [Background] Peet J. Evaluation of the Safety and Efficacy of Hybrid Fractional 2940 nm and 1470 nm Lasers for Treatment of Vaginal Tissue: Pilot Study. [White paper].
- [Derived] Ippolito GM, Crescenze IM, Sitto H, Palanjian RR, Raza D, Barboglio Romo P, Wallace SA, Orozco Leal G, Clemens JQ, Dahm P, Gupta P. Vaginal lasers for treating stress urinary incontinence in women. Cochrane Database Syst Rev. 2025 Jul 25;7(7):CD013643. doi: 10.1002/14651858.CD013643.pub2. PMID 40709601

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited via flyers placed on the UT Southwestern Campus until recruitment concluded in 2020. The first participant was enrolled on June 15, 2018.
Pre-assignment Details: Of the 52 patients enrolled, 5 were screen failures. Hence, total 47 participants were assigned to the interventions. The Placebo Arms (DiVa Sham and IntraGen Sham) are combined here into one Placebo arm since this is how the data was assessed. The Dual Group includes all the Placebo arm participants who initially received 3 placebo treatments and then received 3 dual treatments (DIVA/IntraGen). All subjects assigned to each of the interventions didn't receive treatment between 3-6 months.
Groups:
- Hybrid Fractional Laser (HFL) Group: Patients randomized into the DiVA treatment group will receive treatment per DiVA protocol. Patients will have a total of 3 treatments, space 1 month apart. Each treatment will last approximately 10 minutes. Prior to treatment, the Zimmern probe will be used to measure vaginal wall elasticity and a 0.33mm biopsy will be taken. At each visit, the Zimmern probe will be used. Biopsies will be taken 3 months after final treatment.
  DiVA: DiVA device utilizes a hybrid fractional laser technology in a wand hand piece. The hand piece is covered by a single use strengthened quartz dilator that allows the hand piece to rotate and provide treatment in a uniform manner.
- Radiofrequency (RF) Group: Patients will undergo treatment with radiofrequency device, using the device's standard protocol. Patients will have 3 treatments space one month apart. Each treatment will be a total of 20 minutes for internal treatment only. Prior to treatment, the Zimmern probe will be used to measure vaginal wall elasticity and a 0.33mm biopsy will be taken. At each visit, the Zimmern probe will be used. Biopsies will be taken 3 months after final treatment.
  IntraGen RF: IntraGen is a radiofrequency vaginal rejuvenation device FDA approved for use in dermatological and general surgical procedures for electrocoagulation and hemostasis. The hand piece is a disposable monopolar applicator that is used to apply energy internally and externally.
- Placebo Arm: Participants from the DiVa Sham Group and Intragen Sham Group combined DiVa Placebo: patients will undergo a three-part placebo treatment, spaced 1 month apart (+/- 10 days) of the vulvovaginal area. The vaginal HFL handpiece will be inserted into the vaginal canal but sub-therapeutic energy will not be delivered to the tissue.
  IntraGen Placebo: patients will undergo a three-part placebo treatment, space 1 month apart (+/- 10 days) of the vulvovaginal area. This will be achieved through application of the probe, but with applying sub-therapeutic energy to the tissue.
- Dual (HFL & RF) Group: Patients previously randomized into the DiVA Sham and IntraGen Sham groups will be placed in the Dual Treatment group. Patients will have a total of 3 dual treatments, spaced 1 month apart. Each treatment will last approximately 20 minutes. Prior to dual treatments, the Zimmern probe will be used to measure vaginal wall elasticity and a 0.33mm biopsy will be taken. At each visit, the Zimmern probe will be used. Biopsies will be taken at follow up visits.
  DiVA: DiVA device utilizes a hybrid fractional laser technology in a wand hand piece. The hand piece is covered by a single use strengthened quartz dilator that allows the hand piece to rotate and provide treatment in a uniform manner.
  IntraGen RF: IntraGen is a radiofrequency vaginal rejuvenation device FDA approved for use in dermatological and general surgical procedures for electrocoagulation and hemostasis. The hand piece is a disposable monopolar applicator that is used to apply energy internally and externally.
Period: Initial Intervention (1 to 3 Months)
Arm/Group | Hybrid Fractional Laser (HFL) Group | Radiofrequency (RF) Group | Placebo Arm | Dual (HFL & RF) Group
Started | 12 | 12 | 23 | 0
Completed | 9 | 8 | 14 | 0
Not Completed | 3 | 4 | 9 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 3 | 0
Not completed — Physician Decision | 2 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 2 | 5 | 0
Period: Dual Intervention (6 to 8 Months)
Arm/Group | Hybrid Fractional Laser (HFL) Group | Radiofrequency (RF) Group | Placebo Arm | Dual (HFL & RF) Group
Started | 0 | 0 | 0 | 14
Completed | 0 | 0 | 0 | 14
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Placebo Arms (DiVa Sham and IntraGen Sham) are combined here into one Placebo arm since this is how the data was assessed unlike how it was initially listed in the protocol. The Dual Group includes all the Placebo arm participants who initially received 3 placebo treatments and then received 3 dual treatments (DIVA/IntraGen)
Groups:
- Hybrid Fractional Laser (HFL) Group: Patients randomized into this DiVA treatment group will receive treatment per DiVA protocol. Patients will have a total of 3 treatments, space 1 month apart. Each treatment will last approximately 10 minutes. Prior to treatment, the Zimmern probe will be used to measure vaginal wall elasticity and a 0.33mm biopsy will be taken. At each visit, the Zimmern probe will be used. Biopsies will be taken 3 months after final treatment.
- Radiofrequency (RF) Group: Patients will undergo treatment with radiofrequency device, using the device's standard protocol. Patients will have 3 treatments space one month apart. Each treatment will be a total of 20 minutes for internal treatment only. Prior to treatment, the Zimmern probe will be used to measure vaginal wall elasticity and a 0.33mm biopsy will be taken. At each visit, the Zimmern probe will be used. Biopsies will be taken 3 months after final treatment.
- Placebo Group: Participants from the DiVa Sham Group and Intragen Sham Group combined
  DiVa Placebo: patients will undergo a three-part placebo treatment, spaced 1 month apart (+/- 10 days) of the vulvovaginal area. The vaginal HFL handpiece will be inserted into the vaginal canal but sub-therapeutic energy will not be delivered to the tissue.
  IntraGen Placebo: patients will undergo a three-part placebo treatment, space 1 month apart (+/- 10 days) of the vulvovaginal area. This will be achieved through application of the probe, but with applying sub-therapeutic energy to the tissue.
- Dual (HFL & RF) Group: Patients previously randomized into the DiVA Sham and IntraGen Sham groups will be placed in the Dual Treatment group. Patients will have a total of 3 dual treatments, spaced 1 month apart. Each treatment will last approximately 20 minutes. Prior to dual treatments, the Zimmern probe will be used to measure vaginal wall elasticity and a 0.33mm biopsy will be taken. At each visit, the Zimmern probe will be used. Biopsies will be taken at follow up visits.
- Total: Total of all reporting groups
Arm/Group | Hybrid Fractional Laser (HFL) Group | Radiofrequency (RF) Group | Placebo Group | Dual (HFL & RF) Group | Total
Number analyzed (Participants) | 12 | 12 | 23 | 14 | 61
Age, Categorical [Count of Participants; unit: Participants] — Population: During Initial intervention period there were 0 participants in the dual group. During the dual intervention period there were 14 participants included that were all from the placebo arm who underwent dual intervention and thus were analyzed.
  Participants
    Initial Intervention: number analyzed (Participants) | 12 | 12 | 23 | 0 | 47
    Initial Intervention: <=18 years | 0 | 0 | 0 | 0 | 0
    Initial Intervention: Between 18 and 65 years | 12 | 12 | 23 | 0 | 47
    Initial Intervention: >=65 years | 0 | 0 | 0 | 0 | 0
    Dual Intervention: number analyzed (Participants) | 0 | 0 | 0 | 14 | 14
    Dual Intervention: <=18 years | 0 | 0 | 0 | 0 | 0
    Dual Intervention: Between 18 and 65 years | 0 | 0 | 0 | 14 | 14
    Dual Intervention: >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: During Initial intervention period there were 0 participants in the dual group. During the dual intervention period there were 14 participants included that were all from the placebo arm who underwent dual intervention and thus were analyzed.
  Participants
    Initial Intervention: number analyzed (Participants) | 12 | 12 | 23 | 0 | 47
    Initial Intervention: Female | 12 | 12 | 23 | 0 | 47
    Initial Intervention: Male | 0 | 0 | 0 | 0 | 0
    Dual Intervention: number analyzed (Participants) | 0 | 0 | 0 | 14 | 14
    Dual Intervention: Female | 0 | 0 | 0 | 14 | 14
    Dual Intervention: Male | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Total participants who enrolled and were assigned to the interventions have been included here. Population: During Initial intervention period there were 0 participants in the dual group. During the dual intervention period there were 14 participants included that were all from the placebo arm who underwent dual intervention and thus were analyzed.
  Participants
    Initial Intervention: number analyzed (Participants) | 12 | 12 | 23 | 0 | 47
    Initial Intervention: Caucasian | 5 | 9 | 15 | 0 | 29
    Initial Intervention: Hispanic | 1 | 1 | 2 | 0 | 4
    Initial Intervention: Black or African American | 6 | 2 | 5 | 0 | 13
    Initial Intervention: Caucasian / Hispanic | 0 | 0 | 1 | 0 | 1
    Dual Intervention: number analyzed (Participants) | 0 | 0 | 0 | 14 | 14
    Dual Intervention: Caucasian | 0 | 0 | 0 | 8 | 8
    Dual Intervention: Hispanic | 0 | 0 | 0 | 1 | 1
    Dual Intervention: Black or African American | 0 | 0 | 0 | 4 | 4
    Dual Intervention: Caucasian / Hispanic | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Vulvovaginal Symptoms Questionnaire
Description: VSQ is a 21-item validated survey designed to assess postmenopausal quality-of-life parameters, namely vulvovaginal symptoms, emotions, life and sexual impact.
  Min: 0; Max: 21 Higher score would indicate greater number of symptoms.
Time Frame: Baseline, 3 Month Post- treatments and 6 Month Post Treatments
Population: Subjects originally in DIVA sham and IntraGen Sham arms were combined to create the dual treatment group- these subjects initially received 3 placebo treatments and then received 3 dual treatments (DIVA/IntraGen).
  Our data was not collected at the 6 Month time point for the placebo arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hybrid Fractional Laser (HFL) Group | Radiofrequency (RF) Group | Placebo Arm | Dual (HFL & RF) Group
Number analyzed (Participants) | 9 | 8 | 14 | 14
score on a scale
  Baseline | 8 (5.5) | 7.88 (5.49) | 5.93 (4.67) | 5.93 (4.67)
  3 Month Post Treatment | 3.22 (2.77) | 5 (6.12) | 3 (3.46) | 1.86 (2.51)
  6 Month Post Treatment: number analyzed (Participants) | 9 | 8 | 0 | 14
  6 Month Post Treatment | 3.43 (3.87) | 2.33 (4.41) |  | 1.7 (2.36)

2. Primary Outcome: Vaginal Laxity Questionnaire
Description: The VLQ is a Likert scale with seven responses regarding self-reported vaginal laxity; answer option range from "Very Loose" to "Very Tight".
  Min: 1; Max: 7 A higher score would indicate "Very Tight" response provided by the subject.
Time Frame: Baseline, 3 Months Post Treatments and 6 Months Post Treatments
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hybrid Fractional Laser (HFL) Group | Radiofrequency (RF) Group | Placebo Arm | Dual (HFL & RF) Group
Number analyzed (Participants) | 9 | 8 | 14 | 14
score on a scale
  Baseline | 3.57 (2.51) | 3.67 (2.25) | 2.79 (1.93) | 2.79 (1.93)
  3 Months Post Treatment | 4.44 (1.74) | 3.75 (2.19) | 3.5 (1.74) | 3.93 (1.82)
  6 Months Post Treatment: number analyzed (Participants) | 9 | 8 | 0 | 14
  6 Months Post Treatment | 3.83 (1.72) | 4.5 (1.38) |  | 4.2 (1.4)

3. Secondary Outcome: Perceived Changes in Vaginal Laxity as Measured by Zimmern Probe at 3 Months Post Treatment
Description: Perceived changes in vaginal laxity is measured by Zimmern probe which measures vaginal wall elasticity.
Time Frame: Baseline and 3 Months Post Treatment
Population: Subjects originally in DIVA sham and IntraGen Sham arms were combined to create the dual treatment group- these subjects initially received 3 placebo treatments and then received 3 dual treatments (DIVA/IntraGen). We were unable to collect data for some of the participants who were assigned to each of these arms due to an equipment malfunction and hence these subjects were not included in this analysis.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Hybrid Fractional Laser (HFL) Group | Radiofrequency (RF) Group | Placebo Arm | Dual (HFL & RF) Group
Number analyzed (Participants) | 1 | 5 | 8 | 6
mmHg | 0.44 (NA) — Only 1 participant was analyzed | 0.78 (1.3) | 0.7 (2.47) | 0.36 (1.33)

4. Secondary Outcome: Perceived Changes in Vaginal Laxity as Measured by Zimmern Probe at 6 Months Post Treatment
Description: Perceived changes in vaginal laxity is measured by Zimmern probe which measures vaginal wall elasticity.
Time Frame: Baseline and 6 Months Post Treatment
Population: Collected data were not considered valid due to an equipment malfunction.
Arm/Group | Hybrid Fractional Laser (HFL) Group | Radiofrequency (RF) Group | Placebo Arm | Dual (HFL & RF) Group
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: Urogenital Distress Short Form (UDI-6)
Description: UDI-6 measures multiple domains to assess for presence and severity of physical symptoms such as frequency in urination, urine leakage and pain/discomfort.
  Min: 0; Max: 100 Higher score would indicate a higher disability
Time Frame: Baseline, 3 Months Post Treatments and 6 Months Post Treatments
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hybrid Fractional Laser (HFL) Group | Radiofrequency (RF) Group | Placebo Arm | Dual (HFL & RF) Group
Number analyzed (Participants) | 9 | 8 | 14 | 14
score on a scale
  Baseline | 36.11 (17.92) | 34.38 (24.37) | 28.15 (23.23) | 28.15 (23.23)
  3 Month Post Treatment | 25.65 (18.93) | 41.15 (31.61) | 27.14 (23.11) | 21.13 (23.2)
  6 Month Post Treatment: number analyzed (Participants) | 9 | 8 | 0 | 14
  6 Month Post Treatment | 25.69 (21.8) | 23.61 (20.18) |  | 24.63 (19.16)

6. Secondary Outcome: Incontinence Impact Questionnaire Short Form (IIQ-7)
Description: The Incontinence Impact Questionnaire assesses the impact and extent of incontinence on patients' everyday lives.
  Min: 0; Max: 100 Higher scores corresponds to greater degree of disability.
Time Frame: Baseline, 3 Months Post Treatments and 6 Months Post Treatments
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hybrid Fractional Laser (HFL) Group | Radiofrequency (RF) Group | Placebo Arm | Dual (HFL & RF) Group
Number analyzed (Participants) | 9 | 8 | 14 | 14
score on a scale
  Baseline | 22.75 (18.1) | 22.02 (29.01) | 10.2 (17) | 10.2 (17)
  3 Month Post Treatment | 7.41 (12.62) | 11.31 (13.21) | 15.98 (32.33) | 8.16 (20.24)
  6 Month Post Treatment: number analyzed (Participants) | 9 | 8 | 0 | 14
  6 Month Post Treatment | 11.9 (14.04) | 10.32 (18.42) |  | 10.48 (31.49)

7. Secondary Outcome: Female Sexual Function Index (FSFI)
Description: The FSFI is a 19-item validated questionnaire that assesses several domains of sexual function including, desire, arousal, lubrication, orgasm, satisfaction and pain.
  Min: 2; Max: 36 Higher scores indicate fewer symptoms and greater sexual satisfaction.
Time Frame: Baseline, 3 Months Post Treatments and 6 Months Post Treatments
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hybrid Fractional Laser (HFL) Group | Radiofrequency (RF) Group | Placebo Arm | Dual (HFL & RF) Group
Number analyzed (Participants) | 9 | 8 | 14 | 14
score on a scale
  Baseline | 14.96 (9.23) | 15.69 (10.34) | 15.98 (10.04) | 16.09 (9.62)
  3 Months Post Treatments | 21.38 (11.62) | 18.73 (12.72) | 17.28 (10.98) | 20.67 (10.88)
  6 Months Post Treatments: number analyzed (Participants) | 9 | 8 | 0 | 14
  6 Months Post Treatments | 18.2 (12.33) | 21.7 (14.01) |  | 24.19 (11.06)

8. Secondary Outcome: Gene Expression- Col1A1 as Measured by Fold Change
Description: Biopsies taken of the anterior vaginal wall will be analyzed for gene expression
  Fold change= sample/average of the baseline
Time Frame: Baseline and 3 Months Post Treatments
Population: Study staff was unable to collect a biopsy sample during all visits.
  Subjects originally in DIVA sham and IntraGen Sham arms were combined to create the dual treatment group- these subjects initially received 3 placebo treatments and then received 3 dual treatments (DIVA/IntraGen).
Measure: Mean (Standard Error); unit: fold change
Arm/Group | Hybrid Fractional Laser (HFL) Group | Radiofrequency (RF) Group | Placebo Arm | Dual (HFL & RF) Group
Number analyzed (Participants) | 9 | 8 | 23 | 14
fold change | 0.67 (0.32) | 0.48 (0.24) | 1 (0.25) | 0.95 (0.26)

9. Secondary Outcome: Gene Expression- Col3A1 as Measured by Fold Change
Description: as for outcome 8
Time Frame: Baseline and 3 Months Post Treatments
Population: as for outcome 8
Measure: Mean (Standard Error); unit: fold change
Groups:
- Placebo Arm: Participants from the DiVa Sham Group and Intragen Sham Group combined DiVa Placebo: patients will undergo a three-part placebo treatment, spaced 1 month apart (+/- 10 days) of the vulvovaginal area. The vaginal HFL handpiece will be inserted into the vaginal canal but sub-therapeutic energy will not be delivered to the tissue.
  IntraGen Placebo: patients will undergo a three-part placebo treatment, space 1 month apart (+/- 10 days) of the vulvovaginal area. This will be achieved through application of the probe, but with applying sub-therapeutic en
Arm/Group | Hybrid Fractional Laser (HFL) Group | Radiofrequency (RF) Group | Placebo Arm | Dual (HFL & RF) Group
Number analyzed (Participants) | 9 | 8 | 23 | 14
fold change | 0.95 (0.41) | 0.82 (0.55) | 1 (0.35) | 1.23 (0.25)

10. Secondary Outcome: Gene Expression- ELN as Measured by Fold Change
Description: as for outcome 8
Time Frame: Baseline and 3 Months Post Treatments
Population: as for outcome 8
Measure: Mean (Standard Error); unit: fold change
Groups:
- Placebo Group: Participants from the DiVa Sham Group and Intragen Sham Group combined DiVa Placebo: patients will undergo a three-part placebo treatment, spaced 1 month apart (+/- 10 days) of the vulvovaginal area. The vaginal HFL handpiece will be inserted into the vaginal canal but sub-therapeutic energy will not be delivered to the tissue.
  IntraGen Placebo: patients will undergo a three-part placebo treatment, space 1 month apart (+/- 10 days) of the vulvovaginal area. This will be achieved through application of the probe, but with applying sub-therapeutic en
Arm/Group | Hybrid Fractional Laser (HFL) Group | Radiofrequency (RF) Group | Placebo Group | Dual (HFL & RF) Group
Number analyzed (Participants) | 9 | 8 | 23 | 14
fold change | 0.40 (0.18) | 0.33 (0.20) | 1 (0.16) | 0.79 (0.15)

11. Secondary Outcome: Gene Expression- LOX as Measured by Fold Change
Description: as for outcome 8
Time Frame: Baseline and 3 Months Post Treatments
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: fold change
Arm/Group | Hybrid Fractional Laser (HFL) Group | Radiofrequency (RF) Group | Placebo Arm | Dual (HFL & RF) Group
Number analyzed (Participants) | 9 | 8 | 23 | 14
fold change | 2.72 (1.71) | 0.75 (.28) | 1 (0.16) | 0.95 (0.17)

ADVERSE EVENTS:
Time Frame: 15 months
Arm/Group | Hybrid Fractional Laser (HFL) Group | Radiofrequency (RF) Group | Placebo Arm | Dual (HFL & RF) Group
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/23 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/23 | 0/14
Other Adverse Events (participants affected / at risk) | 7/12 | 4/12 | 6/23 | 6/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Hybrid Fractional Laser (HFL) Group (N=12) | Radiofrequency (RF) Group (N=12) | Placebo Arm (N=23) | Dual (HFL & RF) Group (N=14)
Vaginal Odor/Itching/Spotting (Reproductive system and breast disorders) | 1 | 0 | 1 | 5
UTI/Yeast Infection (Reproductive system and breast disorders) | 0 | 2 | 2 | 0
Urine Leakage (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Abdominal Discomfort (Reproductive system and breast disorders) | 0 | 0 | 1 | 1
Vaginal perspiration (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Other (Reproductive system and breast disorders) | 7 | 4 | 5 | 1 — Symptoms were unrelated to study arms/treatments.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-21): https://cdn.clinicaltrials.gov/large-docs/50/NCT03316950/Prot_SAP_001.pdf